CLINICAL TRIAL: NCT03796156
Title: Aspirin to Target Arterial Events in Chronic Kidney Disease
Acronym: ATTACK
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southampton (Other)
Collaborators: University of Nottingham (Other); University of Warwick (Other); Nottingham University Hospitals NHS Trust (Other); East Kent Hospitals University NHS Foundation Trust (Other Government); University of Durham (Other); Epsom and St Helier University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 31844
Record Dates: First submitted 2018-12-20; First posted 2019-01-08 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Chronic Kidney Diseases; Cardiovascular Diseases; Bleeding
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases; Hemorrhage | interventions — Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Adjudication of outcomes blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin (Experimental): 75mg of non enteric coated or dispersible aspirin once daily added to usual medications
  Interventions: Drug: Aspirin
- Usual care (No Intervention): Usual medications only

INTERVENTIONS:
Drug: Aspirin — 75mg low dose non enteric coated or dispersible
  Arms: Aspirin

SUMMARY:
This study aims to find out whether people with chronic kidney disease [CKD] should take low dose aspirin to reduce the risk of first heart attack or stroke (cardiovascular disease [CVD]). CKD is common and is associated with an increased risk of CVD.

CVD is caused by small blood clots and aspirin thins the blood to reduce the risk of such clots developing but it also increases the risk of bleeding.

Aspirin is recommended to prevent further CVD in people who have already had a first CVD event (so called secondary prevention). Here the investigators want to study the use of aspirin as primary prevention in people with CKD who have not had a CVD to prevent the first event, to assess whether the potential benefits exceed the risks.

Eligible patients will be recruited from their United Kingdom (UK) general practices and allocated by chance to be prescribed once daily low dose aspirin or usual care only. Follow-up will be for several years both electronically (for general practice, hospital and mortality data) and by annual questionnaires to ascertain CVD and bleeding events.

DETAILED DESCRIPTION:
Aim To test the hypothesis that the addition of 75mg aspirin once daily to usual care reduces the risk of major vascular events in patients with chronic kidney disease (CKD) who do not have pre-existing cardiovascular disease (CVD)

Design Open label, multi-centre randomised controlled trial

Setting UK general practices

Sample size 25,210 patients (12,605 per arm). A total of 1,827 major vascular events overall are required.

Eligibility Inclusion Criteria

1. Males and females aged 18 years and over at the date of screening
2. Subjects with CKD (reduced eGFR and/or albuminuria) defined as: • estimated glomerular filtration rate [eGFR] <60mL/min/1.73m2 for at least 90 days, and/or • kidney disease code on the GP electronic patient AND most recent eGFR in CKD-defining range (<60mL/min/1.73m2), and/or • albuminuria or proteinuria (defined as urine albumin:creatinine ratio [ACR] ≥3mg/mmol, and/or urine protein:creatinine ratio [PCR] ≥15mg/mmol, and/or +protein or greater on reagent strip)
3. Subjects who are willing to give permission for their paper and electronic medical records to be accessed by trial investigators
4. Subjects who are willing to be contacted and interviewed by trial investigators
5. Subjects who can communicate well with the investigator or designee, understand the requirements of the study and understand and sign the written informed consent

Exclusion Criteria

1. Subjects with CKD eGFR category 5
2. Subjects with pre-existing cardiovascular disease (angina, myocardial infarction, stroke, transient ischaemic attack (TIA), significant peripheral vascular disease, coronary or peripheral revascularisation for atherosclerotic disease)
3. Subjects with a current pre-existing condition associated with increased risk of bleeding other than CKD
4. Subjects currently prescribed anticoagulants or antiplatelet agent, or taking over the counter (OTC) aspirin continuously
5. Subjects who are currently and regularly taking other drugs with a potentially serious interaction with aspirin
6. Subjects with a known allergy to aspirin or definite previous clinically important adverse reaction
7. Subjects with poorly controlled hypertension (systolic blood pressure [BP] ≥180 mmHg and/or diastolic BP ≥105 mmHg)
8. Subjects with other conditions which in the opinion of their General Practitioner (GP) would preclude prescription of aspirin in routine clinical practice, for example significant anaemia or thrombocytopenia.
9. Subjects who are pregnant or likely to become pregnant during the study period
10. Subjects with malignancy that is life-threatening or likely to limit prognosis, other life-threatening co-morbidity, or terminal illness
11. Subjects whose behaviour or lifestyle would render them less likely to comply with study medication
12. Subjects in prison
13. Subjects currently participating in another clinical trial of an investigational medicinal product or who have taken part in such a trial in the last three months (Covid-19 vaccine studies are acceptable)

Interventions Suitable participants will be randomised to receive: 75mg non-enteric coated or dispersible aspirin once daily in addition to their usual medication; or no additional treatment and avoidance of aspirin.

Duration The trial will continue until at least 1,827 adjudicated primary endpoint events (major vascular events) have occurred, or before if the trial is discontinued after the internal pilot or for any other reason. It is anticipated that at least 6 years of recruitment (taking account a recruitment pause for the Covid-19 pandemic) and 2.5 years of follow-up will be required to complete the trial.

Randomisation and blinding Eligible participants, based on results of routine blood and urine tests at screening, will be randomised (open label randomisation) 1:1 to general practitioner (GP) prescription of aspirin vs. no prescription, stratified by age, diabetes and CKD severity.

Follow-up Data on potential CVD and bleeding outcomes will be collected electronically from GP records and national hospitalisation and mortality records. Adjudication panels (for CVD and for bleeding) will asses the information blind to allocation.

Patients will complete an annual quality of life questionnaire (EQ5D).

Outcomes. Primary outcome measure

Time to first major vascular event from the date of randomisation. A major vascular event is defined as a primary composite outcome of non-fatal myocardial infarction (MI), non-fatal stroke and cardiovascular death (excluding confirmed intracranial haemorrhage and other fatal cardiovascular haemorrhage).

Secondary outcome measures (all time to event except quality of life)

Efficacy

1. Death from any cause
2. Composite outcome of major vascular event or revascularisation (coronary and non-coronary)
3. Individual components of the primary composite endpoint
4. Health-related quality of life

Safety

1. Composite outcome of intracranial haemorrhage (fatal and non-fatal), fatal extracranial haemorrhage and non-fatal major extracranial haemorrhage (adjudicated)
2. Fatal and non-fatal (reported individually and as a composite) intracranial haemorrhage comprising: i) primary haemorrhagic stroke (to distinguish from haemorrhagic transformation of ischaemic stroke); ii) other intracranial haemorrhage (adjudicated). Intra-cranial haemorrhage will be sub-categorised as traumatic or non-traumatic.
3. Fatal and non-fatal (reported individually and as a composite) major extracranial haemorrhage: i) upper gastrointestinal; ii) lower gastrointestinal; iii) sight-threatening ocular; iv) multiple trauma; v) other (adjudicated).
4. Clinically relevant non-major bleeding if hospitalised (adjudicated).
5. Composite outcome of fatal and non-fatal major extracranial haemorrhage and clinically relevant non-major bleeding (if hospitalised).

Tertiary (exploratory) outcome measures (all time to event except hospitalisation)

1. Transient ischaemic attack
2. Unplanned hospitalisation
3. Hospitalisation with heart failure
4. New diagnosis of cancer (colorectal/other)
5. Death due to cancer (where cancer is the underlying cause of death)
6. CKD progression
7. New diagnosis of dementia
8. Major non-traumatic lower limb amputation

Statistical methods The primary outcome measure of time to first major vascular event will be analysed for the intention-to-treat (ITT) population. Deaths from other causes (including fatal bleeding) will be treated as competing events. Patients who do not experience a major vascular event will be censored at the date of last follow-up.

All primary, secondary and tertiary time to event outcomes will be described using Kaplan-Meier curves or Cumulative Hazard plots for time to event outcomes involving competing risks for the ITT population. Analyses of time to event outcomes will be performed using Cox proportional hazards models or Competing Risk regression models, both unadjusted and adjusted for stratification factors: age, diabetes and CKD severity.

The adjusted Competing Risk regression model for time to first major vascular event, with deaths from other causes (including fatal bleeding) treated as competing events, and patients who do not experience a major vascular event censored, will form the primary endpoint analysis model.

Other secondary and tertiary endpoints will be assessed by arm using summary statistics (e.g. Pearson's χ² tests) in the ITT population.

The amount of missing data and reasons for the incompleteness will be explored and presented overall i.e. not by group. If the amount of missing data is deemed too high and if appropriate (i.e. assuming the missing data is either missing at random [MAR] or missing completely at random [MCAR] and censoring assumed to be non-informative), multiple imputation will be performed accordingly, for which all covariates included in the multivariable model, together with the censoring/event indicator and the cumulative baseline hazard will be included in the multiple imputation model.

Health economic analysis will also be undertaken.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 years and over at the date of screening
* .Subjects with CKD (reduced eGFR and/or albuminuria) defined as: • estimated glomerular filtration rate [eGFR] <60mL/min/1.73m2 for at least 90 days, and/or • kidney disease code on the GP electronic patient AND most recent eGFR in CKD-defining range (<60mL/min/1.73m2), and/or • albuminuria or proteinuria (defined as urine albumin:creatinine ratio [ACR] ≥3mg/mmol, and/or urine protein:creatinine ratio [PCR] ≥15mg/mmol, and/or +protein or greater on reagent strip)
* Subjects who are willing to give permission for their paper and electronic medical records to be accessed by trial investigators
* Subjects who are willing to be contacted and interviewed by trial investigators
* Subjects who can communicate well with the investigator or designee, understand the requirements of the study and understand and sign the written informed consent

Exclusion Criteria

* Subjects with CKD GFR category 5
* Subjects with pre-existing cardiovascular disease (angina, myocardial infarction, stroke, transient ischaemic attack (TIA), significant peripheral vascular disease, coronary or peripheral revascularisation for atherosclerotic disease)
* Subjects with a current pre-existing condition associated with increased risk of bleeding other than CKD
* Subjects currently prescribed anticoagulants or antiplatelet agent, or taking over the counter (OTC) aspirin continuously
* Subjects who are currently and regularly taking other drugs with a potentially serious interaction with aspirin
* Subjects with a known allergy to aspirin or definite previous clinically important adverse reaction
* Subjects with poorly controlled hypertension (systolic blood pressure [BP] ≥180 mmHg and/or diastolic BP ≥105 mmHg)
* . Subjects with other conditions which in the opinion of their General Practitioner (GP) would preclude prescription of aspirin in routine clinical practice, for example significant anaemia or thrombocytopenia
* Subjects who are pregnant or likely to become pregnant during the study period
* Subjects with malignancy that is life-threatening or likely to limit prognosis, other life-threatening co-morbidity, or terminal illness
* Subjects whose behaviour or lifestyle would render them less likely to comply with study medication
* Subjects in prison
* Subjects currently participating in another clinical trial of an investigational medicinal product or who have taken part in such a trial in the last three months (Covid-19 vaccine studies are acceptable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25210 (Estimated)
Dates: Start 2019-02-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a Major vascular event: Composite outcome of non-fatal myocardial infarction, non-fatal stroke and cardiovascular death (excluding confirmed intracranial haemorrhage and other fatal cardiovascular haemorrhage) | Over average 4 years follow-up
  Acute MI defined according to the Third Universal Definition of myocardial infarction (MI).
  Acute stroke defined in accordance with the World Health Organization (WHO) definition as "rapidly developing clinical signs of focal (or global) disturbance of cerebral function, with symptoms lasting 24 hours or longer, with no apparent cause other than of vascular origin". This excludes cases of primary cerebral tumour, cerebral metastasis, subdural haematoma, post-seizure palsy, brain trauma and TIA. Haemorrhagic stroke (fatal and non-fatal) including intracerebral haemorrhage and SAH which has been confirmed on appropriate imaging is excluded from the primary composite endpoint and included within the secondary endpoints.

SECONDARY OUTCOMES:
Number of participants dying from any cause | Average 4 years follow-up
  Death from any cause
Number of participants with major vascular events plus revascularisation | Average 4 years follow-up
  Primary outcome plus coronary and non coronary arterial revascularisation. It will include open and percutaneous coronary and non-coronary (including carotid, aortic and limb) procedures (as defined in Office of Population Censuses and Surveys OPCS-4 procedure codes) and will be ascertained from Hospital Episode Statistics (HES) data.
Number of participants with Non-fatal myocardial infarction | Average 4 years follow-up
  Non-fatal myocardial infarction. Acute MI defined according to the Third Universal Definition of myocardial infarction (MI).
Health-related quality of life, mean utility score | Average 4 years follow-up
  Euroqol EQ-5D utility score derived from 5 states (scoring 1-5) converted to utility values using UK general population set
Number of participants with intra-cranial haemorrhage, fatal and non fatal major extra cranial haemorrhage | Average 4 years follow-up
  Intra-cranial haemorrhage includes intracerebral haemorrhage, subarachnoid haemorrhage, subdural haemorrhage, and extradural haemorrhage.
  Extra-cranial haemorrhage is:
  * Fatal bleeding, or
  * Symptomatic bleeding in a critical area or organ, such as intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome, or
  * Bleeding that leads to the transfusion of two or more units of whole blood or red cells
  In particular, to be classified as major, bleeds in a critical area or organ should:
  * Be associated with a symptomatic clinical presentation (not following an incidental finding)
  * Be the cause of the symptoms
Number of participants with Fatal and non-fatal intra-cranial haemorrhage | Average 4 years follow-up
  Fatal and non-fatal intra-cranial haemorrhage as above It comprises primary haemorrhagic stroke(to distinguish from haemorrhagic transformation of ischaemic stroke) ii)other intra-cranial haemorrhage (adjudicated). Intra-cranial haemorrhage will be sub categorised as traumatic and non-traumatic.
Number of participants with Fatal and non-fatal major extra-cranial haemorrhage | Average 4 years follow-up
  Fatal and non-fatal major extra-cranial haemorrhage as above. Categorised as i) upper-gastro-intestinal ii) lower gastro-intestinal iii) sight threatening ocular iv)multiple trauma v) other
Number of participants with Clinically relevant non major bleeding (hospitalised) | Average 4 years follow-up
  Defined in accordance with the International Society on Thrombosis and Haemostasis (ISTH) as any sign or symptom of haemorrhage (e.g. more bleeding than would be expected for a clinical circumstance, including bleeding found by imaging alone) that does not fit the criteria for the ISTH definition of major bleeding but does meet at least one of the following criteria:
  • Leading to hospitalisation
  This definition excludes all minor bleeding episodes that lead to medical evaluation involving direct patient contact.
Number of participants with Non-fatal stroke | Average 4 years follow-up
  Non-fatal stroke excluding confirmed intracranial haemorrhage. Acute stroke defined in accordance with the World Health Organization (WHO) definition as "rapidly developing clinical signs of focal (or global) disturbance of cerebral function, with symptoms lasting 24 hours or longer, with no apparent cause other than of vascular origin". This excludes cases of primary cerebral tumour, cerebral metastasis, subdural haematoma, post-seizure palsy, brain trauma and TIA. Haemorrhagic stroke ( including intracerebral haemorrhage and sub-arachnoid haemorrhage) which has been confirmed on appropriate imaging is excluded.
Number of participants with Cardiovascular death | Average 4 years follow-up
  Cardiovascular death (excluding confirmed intracranial haemorrhage and other fatal cardiovascular haemorrhage).
Number of participants with fatal and non fatal major extra-cranial haemorrhage and clinically relevant non major bleed (if hospitalised) | Average 4 years follow-up
  Definitions above

OTHER OUTCOMES:
Number of participants with transient ischaemic attack | Average 4 years follow-up
  A transient episode of neurological dysfunction caused by focal brain spinal cord or retinal ischemia without acute infarction
Number of Unplanned hospitalisations per participant | Average 4 years follow-up
  Defined as an official admission that is for a duration greater than 24 hours or a minimum of 2 calendar days where exact time of stay is unavailable.
Number of participants with new diagnosis of cancer | Average 4 years follow-up
  Any new cancer diagnosis excluding non melanotic skin cancer
Number of participants with CKD progression | Average 4 years follow-up
  Defined as at least one of:
  * >30% fall in eGFR over two years, or
  * need for renal replacement therapy or 50% decline in eGFR, or
  * new eGFR<15mL/min/1.73m2, or
  * 25% decline in GFR together with a drop in GFR category
Number of participants with new diagnosis of dementia | Average 4 years follow-up
  Coded dementia (ICD, Read) from linked GP and hospital data
Hospitalisation with heart failure | Average 4 years follow-up
  Coded heart failure (ICD) from hospitalisation data
Death due to cancer (where cancer is the underlying cause of death) | Average 4 years follow-up
Major non traumatic lower limb amputation | Average 4 years follow-up
  Below or above knee amputation, coded (ICD) from hospitalisation data

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Gallagher, MD, Principal Investigator — Epsom and St Helier University Hospitals NHS Trust; Paul Roderick, MD, Principal Investigator — University of Southampton
Locations (1):
- Nottingham Digestive Diseases Centre, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gallagher H, Dumbleton J, Maishman T, Whitehead A, Moore MV, Fuat A, Fitzmaurice D, Henderson RA, Lord J, Griffith KE, Stevens P, Taal MW, Stevenson D, Fraser SD, Lown M, Hawkey CJ, Roderick PJ. Aspirin to target arterial events in chronic kidney disease (ATTACK): study protocol for a multicentre, prospective, randomised, open-label, blinded endpoint, parallel group trial of low-dose aspirin vs. standard care for the primary prevention of cardiovascular disease in people with chronic kidney disease. Trials. 2022 Apr 21;23(1):331. doi: 10.1186/s13063-022-06132-z. PMID 35449015
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730